CLINICAL TRIAL: NCT03341260
Title: Effect of Preoperative, Single-dose Diclofenac Potassium on Postoperative Endodontic Pain in Patients With Symptomatic Irreversible Pulpitis: A Double Blind Randomized Controlled Trial
Brief Title: Effect of Preoperative Diclofenac Potassium on Postoperative Endodontic Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amatallah Hussein Nasser Al-Rawhani, Postgraduate Student in Endodontic Department/ Faculty of Oral and Dental Medicine/ Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBC-CU-2016-11-167
Record Dates: First submitted 2017-11-05; First posted 2017-11-14 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Pulpitis - Irreversible
Keywords: Pulpitis, irreversible Pulpitis,; Diclofenac Potassium; Premedication, Preoperative Analgesic; Postoperative pain
MeSH Terms: conditions — Pulpitis; Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: The patients will be randomly divided into 2 groups:
  Experimental group:
  50 mg Diclofenac Potassium to be administered one hour before treatment.
  Control group:
  Placebo to be administered one hour before treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diclofenac Potassium 50mg tab (Experimental): Diclofenac Potassium 50mg tablet to be administered one hour before treatment.
  Interventions: Drug: Diclofenac Potassium 50mg Tab.
- Placebo (Placebo Comparator): Placebo to be administered one hour before treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Potassium 50mg Tab. — A 50 mg tablet of the medication to be taken one hour before initiation of endodontic treatment.
  Arms: Diclofenac Potassium 50mg tab
Drug: Placebo — A placebo will be taken one hour before initiation of endodontic treatment.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of preoperative a single-dose of 50 mg diclofenac potassium on postoperative endodontic pain in mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Patients with moderate-to-severe preoperative pain are selected. Patients receive either a single-dose of 50 mg diclofenac potassium (group A) or a placebo tablet as a control (group B). All patients receive the assigned premedication one hour before single-visit root canal treatment. Postoperative endodontic pain is measured at the following time points: 6 , 12,24,48 h after treatment. The incidence of analgesic intake is also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active pain (moderate-to-severe) in mandibular molars.
* Patients with prolonged response to cold testing and electric pulp tester.
* Patient with the ability to understand and use pain scales.
* Patient with vital coronal pulp tissue on access.
* Patient who accept to enroll to the study.

Exclusion Criteria:

* Patients' allergies or any other contraindication to diclofenac potassium or articaine.
* Pregnant and lactating females.
* Patients having pain medication in the last 6 hours.
* Patient has more than one symptomatic mandibular tooth in the same quadrant.
* Patients with periradicular pathosis and/or radiolucency other than widened periodontal ligaments.
* Patients with active peptic ulcer and gastrointestinal disorders.
* Patients with history of bleeding problems or anticoagulant use within the last month.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Postoperative endodontic pain | Up to 2 days after endodontic treatment
  Pain after completion root canal treatment measured by Heft-parker visual analogue scale.

SECONDARY OUTCOMES:
Analgesic intake | Up to 2 days after endodontic treatment
  The incidence of analgesic intake is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Amatallah H Al-Rawhani, Pos, Principal Investigator — Faculty of Oral and Dental Medicine/ Cairo University.
Locations (1):
- Dentistry Faculty, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elzaki WM, Abubakr NH, Ziada HM, Ibrahim YE. Double-blind Randomized Placebo-controlled Clinical Trial of Efficiency of Nonsteroidal Anti-inflammatory Drugs in the Control of Post-endodontic Pain. J Endod. 2016 Jun;42(6):835-42. doi: 10.1016/j.joen.2016.02.014. Epub 2016 Apr 12. PMID 27080115
- [Background] Metri M, Hegde S, Bhandi S. Effect of pretreatment diclofenac sodium on postendodontic pain: A randomised controlled trial. J Conserv Dent. 2016 Jan-Feb;19(1):7-10. doi: 10.4103/0972-0707.173183. PMID 26957785